CLINICAL TRIAL: NCT00732914
Title: A Phase III Randomized Sequential Open-Label Study to Evaluate the Efficacy and Safety of Sorafenib Followed by Sunitinib Versus Sunitinib Followed by Sorafenib in the Treatment of First-Line Advanced / Metastatic Renal Cell Carcinoma
Brief Title: Sequential Study to Treat Renal Cell Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sponsor GmbH (Other)
Collaborators: iOMEDICO AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09072008-13772; EudraCT 2008-005011-18
Record Dates: First submitted 2008-08-11; First posted 2008-08-12 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Renal Cell Carcinoma
Keywords: Renal Cell Carcinoma; Sunitinib; Sorafenib; Sequential
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sunitinib; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Sunitinib (first-line) followed by Sorafenib (second-line)
  Interventions: Drug: Sunitinib (Sutent)
- 2 (Experimental): Sorafenib (first-line) followed by Sunitinib (second-line)
  Interventions: Drug: Sorafenib (Nexavar)

INTERVENTIONS:
Drug: Sunitinib (Sutent) — Sunitinib 50 mg once daily 4 weeks on, 2 weeks off, and after discontinuation (due to PD or toxicity), followed by sorafenib 400 mg BID
  Arms: 1
Drug: Sorafenib (Nexavar) — Sorafenib 400 mg BID, followed by Sunitinib 50 mg once daily 4 weeks on, 2 weeks off, and after discontinuation (due to PD or toxicity)
  Arms: 2

SUMMARY:
Primary:

To evaluate if progression-free survival from first treatment to progression or death during second-line therapy (total PFS) of sorafenib followed by sunitinib is superior compared to sunitinib followed by sorafenib.

Secondary:

1. Time from first treatment to progression during second-line therapy (total TTP)
2. Time to first-line treatment failure (progression, death, discontinuation due to toxicity) descriptively in each arm
3. PFS in first-line and second-line treatment, descriptively
4. Overall survival, descriptively (data cut-off same as for primary endpoint)
5. Disease Control Rate (DCR); Response rates in first-line and in second-line (CR, PR, SD according to RECIST criteria)
6. Cardiotoxicity analysis by means of echocardiography and NT-pro BNP with an interim analysis after 100 patients of each arm have completed the study
7. Safety and tolerability

DETAILED DESCRIPTION:
The results of three sequential retrospective studies (Sablin et al, ASCO 2007; Dham et al, ASCO 2007; and Tamaskar et al, 2008) support the sequential administration of sorafenib and sunitinib even though these two drugs have an overlap of targets. These results suggest the lack of cross resistance between sorafenib and sunitinib. This study is a sequential, randomized, open-label (1:1), multicenter phase III study starting in first-line of metastatic / advanced RCC using in the experimental arm sorafenib until progression followed by sunitinib and in the control arm sunitinib until progression followed by sorafenib. Sorafenib-patients will switch to sunitinib and vice versa, with a treatment-free period of at least one and up to maximum four weeks after confirmed first-line treatment failure, in order to avoid additive toxicity. In general, the first-line treatment should be continued until progression (RECIST). However, if patients do not tolerate the first-line medication (sorafenib or sunitinib) because of toxicity, they may cross-over to the second-line therapy (sunitinib or sorafenib) despite the lack of progression, if an appropriate attempt according to a specific dose reduction / interruption scheme has been made to cope with the toxicity and try to resume first line therapy, if deemed appropriate with a reduced dose. In case of discontinuation of first-line treatment because of toxicity, patients will be enrolled for the second-line treatment, only after nonhematological toxicity has resolved to grade ≤1 and hematological toxicity to grade ≤2. As an exception, patients who refuse to be treated further with the first-line regimen due to intolerability despite having no progression may be crossed over to the second-line treatment, if they consent and are in general compliance. Any crossover, also without progression, requires a CT scan, which is in this case also considered the baseline scan for the second-line treatment. One cycle is of six weeks duration. Patients will undergo a CT/MRI scan after every second cycle (i.e. after 12 weeks each), which will be evaluated according to RECIST criteria. There will be no continuation of the same study medication beyond progression in both first- or second-line therapy. After the study reached its primary endpoint cut off, i.e. after 194 endpoint events have occurred, clean data for these patients exist and a statistical analysis has been performed data collection will be stopped. After that the trial is terminated and a close out visit will be performed. Remaining patients will be treated outside the study and will be censored in the analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with metastatic / advanced RCC (all histologies), who are not suitable for cytokine therapy and for whom study medication constitutes first-line therapy
2. Age >= 18 ans <= 85years
3. ECOG Performance Status of 0 or 1
4. MSKCC prognostic score, low or intermediate
5. Life expectancy of at least 12 weeks.
6. Subjects with at least one uni-dimensional (for RECIST) measurable lesion. Lesions must be measured by CT/MRI-scan.
7. Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to start of therapy:

   * Hemoglobin >= 9.0 g/dl
   * Absolute neutrophil count (ANC) >= 1,500/mm³
   * Platelet count >= 100,000/μl
   * Total bilirubin <= 1.5 times the upper limit of normal
   * ALT and AST <= 2.5 x upper limit of normal (<= 5 x upper limit of normal for patients with liver involvement of their cancer)
   * Alkaline phosphatase < 4 x upper limit of normal
   * PT-INR/PT < 1.5 x upper limit of normal [Patients who are being therapeutically anticoagulated with an agent such as coumadin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in these parameters exists.]
   * Serum creatinine <= 2 x upper limit of normal.
8. Written Informed Consent

Exclusion Criteria:

1. History of cardiac disease: congestive heart failure >NYHA class 2 or with LVEF at baseline echocardiography < 50%; active CAD (MI more than 6 months prior to study entry is allowed); cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted) or uncontrolled hypertension (defined as blood pressure >= 160 mmHg systolic and/or >= 90 mmHG diastolic on medication).
2. History of HIV infection or chronic hepatitis B or C
3. Active clinically serious infections (> grade 2 NCI-CTC version 3.0)
4. Symptomatic metastatic brain or meningeal tumors (unless the patient is > 6 months from definitive therapy, has a negative imaging study within 4 weeks of study entry and is clinically stable with respect to the tumor at the time of study entry)
5. Patients with seizure disorder requiring medication (such as steroids or anti-epileptics)
6. History of organ allograft
7. Patients with evidence or history of bleeding diathesis
8. untreated hypothyrosis
9. Patients undergoing renal dialysis
10. Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors [Ta, Tis & T1] or any cancer curatively treated > 3 years prior to study entry.
11. Pregnant or breast-feeding patients. Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start of treatment. Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial and 3 months after the completion of trial.
12. Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
13. Any condition that is unstable or could jeopardize the safety of the patient and their compliance in the study
14. Patients unable to swallow oral medications
15. Known allergy to sunitinib or sorafenib or one of its constituents

Excluded therapies and medications, previous and concomitant:

1. Anticancer chemotherapy or immunotherapy during the study or within 4 weeks of study entry.
2. Radiotherapy during study or within 3 weeks of start of study drug. (Palliative radiotherapy will be allowed). Major surgery within 4 weeks of start of study
3. Autologous bone marrow transplant or stem cell rescue within 4 months of study
4. Use of biologic response modifiers, such as G-CSF, within 3 week of study entry.

   [G-CSF and other hematopoietic growth factors may be used in the management of acute toxicity such as febrile neutropenia when clinically indicated or at the discretion of the investigator; however they may not be substituted for a required dose reduction.] [Patients taking chronic erythropoietin are permitted provided no dose adjustment is undertaken within 2 months prior to the study or during the study]
5. Investigational drug therapy outside of this trial during or within 4 weeks of study entry
6. Prior exposure to the study drug.
7. Any St. John's wort containing remedy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2009-01; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
total Progression Free Survival | Last patient last visit (LPLV) to October 2013

SECONDARY OUTCOMES:
Total Time to Progression | Last patient last visit (LPLV) to October 2013
Overall survival | Last patient last visit (LPLV) to October 2013
Disease Control Rate (DCR) | Last patient last visit (LPLV) to October 2013
Cardiotoxicity | after 100 patients of each arm have completed the study

CONTACTS AND LOCATIONS:
Locations (1):
- Urologische Klinik, Mannheim, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Aldin A, Besiroglu B, Adams A, Monsef I, Piechotta V, Tomlinson E, Hornbach C, Dressen N, Goldkuhle M, Maisch P, Dahm P, Heidenreich A, Skoetz N. First-line therapy for adults with advanced renal cell carcinoma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 May 4;5(5):CD013798. doi: 10.1002/14651858.CD013798.pub2. PMID 37146227
- [Derived] Eichelberg C, Vervenne WL, De Santis M, Fischer von Weikersthal L, Goebell PJ, Lerchenmuller C, Zimmermann U, Bos MM, Freier W, Schirrmacher-Memmel S, Staehler M, Pahernik S, Los M, Schenck M, Florcken A, van Arkel C, Hauswald K, Indorf M, Gottstein D, Michel MS. SWITCH: A Randomised, Sequential, Open-label Study to Evaluate the Efficacy and Safety of Sorafenib-sunitinib Versus Sunitinib-sorafenib in the Treatment of Metastatic Renal Cell Cancer. Eur Urol. 2015 Nov;68(5):837-47. doi: 10.1016/j.eururo.2015.04.017. Epub 2015 May 4. PMID 25952317
- [Derived] Calvani N, Morelli F, Leo S, Orlando L, Lombardi L, Gnoni A, Cinefra M, Maiello E, Lorusso V, Cinieri S. Sequential use of sorafenib and sunitinib in advanced renal cell carcinoma: does the order of sequencing matter? Med Oncol. 2012 Sep;29(3):1908-13. doi: 10.1007/s12032-011-0048-0. Epub 2011 Aug 20. PMID 21858552